CLINICAL TRIAL: NCT02703259
Title: Single Dose Preoperative Gabapentin Use in Minimally Invasive Hysterectomy for Acute Pain Management
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 603262
Record Dates: First submitted 2016-02-24; First posted 2016-03-09 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Gabapentin; Acetaminophen; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gabapentin (Active Comparator): As per the enhanced recovery after surgery protocol at our health institution, subject will receive oral medications prior to surgery including acetaminophen, celecoxib, and gabapentin x 1 dose given preoperatively. The number of tablets and capsules will remain identical in both study arms. Medications given include:
  Gabapentin 600 mg (two capsules of gabapetin 300 mg); Acetaminophen 975 mg (three tablets of acetaminophen 325 mg); Celecoxib 400 mg (two capsules of celecoxib 200 mg) = Total 3 tablets, 4 capsules
  Interventions: Drug: Gabapentin; Drug: Acetaminophen; Drug: Celecoxib
- Control (Placebo Comparator): As per the enhanced recovery after surgery protocol at our health institution, subject will receive oral medications prior to surgery including acetaminophen and celecoxib x 1 dose given preoperatively. The number of tablets and capsules will remain identical in both study arms. Medications given include:
  Acetaminophen 975 mg (three tablets of acetaminophen 325 mg); Celecoxib 400 mg (four capsules of celecoxib 100 mg) = Total total 3 tablets, 4 capsules
  Interventions: Drug: Acetaminophen; Drug: Celecoxib

INTERVENTIONS:
Drug: Gabapentin
  Arms: Gabapentin
Drug: Acetaminophen
Drug: Celecoxib

SUMMARY:
The purpose of the investigators' study is to assess the efficacy of a single dose of preoperative gabapentin within an enhanced recovery after surgery protocol in acute postoperative pain reduction for women undergoing a minimally invasive hysterectomy. Participants who consent to participate will be randomized to either a control group without gabapentin or to a study arm and receive gabapentin 600 mg prior to their planned surgery. The investigators will collect data on postoperative narcotic use, subjective pain as rated by a numeric pain scale, in addition to any adverse effects of single dose gabapentin use.

DETAILED DESCRIPTION:
Multimodal postoperative analgesia after a hysterectomy has been mainly based on a combination of nonsteroidal anti-inflammatory drugs and opioids. However, adverse effects including nausea, vomiting, sedation, and pruritus may limit use of opioids. As the side effects are dose related, minimizing opioid exposure may significantly reduce these risks. Thus, there has been an interest in evaluating preemptive as well as post-operative administration of non-opioids. Additional regimens have been suggested to minimize opioid use and its associated adverse effects including injection of local anesthetics, epidural analgesia, and anticonvulsants, such as gabapentin or pregabalin.

Gabapentin, a widely used anticonvulsant used for treatment of neuropathic pain, has recently been suggested to improve postoperative analgesia and reduce opioid requirements. Gabapentin is thought to modulate calcium channels on the presynaptic nociceptive neurons, which in turn modulate or inhibit the release of excitatory neurotransmitters from activated nociceptors. In addition to inhibiting pain transmission, gabapentin may exert an analgesic effect by activating descending inhibitory noradrenergic pathways.

Many studies have demonstrated the safety and efficacy of gabapentin for perioperative use in a variety of procedures across disciplines including thoracotomy, laparoscopic cholecystectomy, tonsillectomy, major orthopedic surgery, cesarean sections, and abdominal hysterectomy. Several randomized trials have evaluated the effects of gabapentin administered preoperatively only as well as given pre- and postoperatively for hysterectomy. In a systematic review of 14 studies conducted between 2004 and 2013, with samples ranging from 40 to 200, investigators identified 8 trials in which gabapentin was administered only preoperatively to reduce pain associated with abdominal hysterectomy surgery. Analysis of those data clearly demonstrates that preemptive gabapentin reduced the postoperative visual analog scale (VAS) pain score by approximately 50% and postoperative use of morphine by approximately 37%. The incidence of pruritus and dry mouth in those receiving preemptive gabapentin appeared similar to those receiving placebo, however there was a higher rate of reported dizziness (not statistically significant) associated with gabapentin. In contrast, multiple postoperative doses of gabapentin in addition to the preoperative dose was found to have no significant effect on VAS scores at 24 hours, thus favoring a single preoperative dose.

Although initial results have been encouraging, uptake of gabapentin in routine clinical use remains limited due to mixed results and variability between gabapentin protocols, including dosing and duration. Christiana Care Health System (CCHS) plans to implement the Enhanced Recovery After Surgery (ERAS) protocol which administers preoperative medications to reduce postoperative pain, including acetaminophen, celecoxib, dexamethasone, and gabapentin. Therefore the aim of this study is to assess the efficacy of a single dose of preoperative gabapentin protocol to reduce acute postoperative pain in women undergoing a minimally invasive hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* undergoing a minimally invasive hysterectomy with surgeons operating within the Christiana Care Health System at the Newark location only.
* at least 18 years of age
* able to swallow tablets or capsules

Exclusion Criteria:

* liver failure
* renal failure
* prior gastric bypass
* gastroparesis
* recent or current regular gabapentin use
* hypersensitivity to gabapentin, acetominophen, or celecoxib
* procedure is converted to laparotomy for any indication. (Mini-laparotomy for specimen removal alone will not be excluded.)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2016-06; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terri Huynh, MD, Principal Investigator — Christiana Care Health Services; Gretchen Makai, MD, Principal Investigator — Christiana Care Health Services
Locations (1):
- Christiana Care Health System, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alayed N, Alghanaim N, Tan X, Tulandi T. Preemptive use of gabapentin in abdominal hysterectomy: a systematic review and meta-analysis. Obstet Gynecol. 2014 Jun;123(6):1221-1229. doi: 10.1097/AOG.0000000000000289. PMID 24807337
- [Background] Clarke H, Bonin RP, Orser BA, Englesakis M, Wijeysundera DN, Katz J. The prevention of chronic postsurgical pain using gabapentin and pregabalin: a combined systematic review and meta-analysis. Anesth Analg. 2012 Aug;115(2):428-42. doi: 10.1213/ANE.0b013e318249d36e. Epub 2012 Mar 13. PMID 22415535
- [Background] Dolin SJ, Cashman JN. Tolerability of acute postoperative pain management: nausea, vomiting, sedation, pruritus, and urinary retention. Evidence from published data. Br J Anaesth. 2005 Nov;95(5):584-91. doi: 10.1093/bja/aei227. Epub 2005 Sep 16. PMID 16169893
- [Background] Schmidt PC, Ruchelli G, Mackey SC, Carroll IR. Perioperative gabapentinoids: choice of agent, dose, timing, and effects on chronic postsurgical pain. Anesthesiology. 2013 Nov;119(5):1215-21. doi: 10.1097/ALN.0b013e3182a9a896. No abstract available. PMID 24051389
- [Background] Straube S, Derry S, Moore RA, Wiffen PJ, McQuay HJ. Single dose oral gabapentin for established acute postoperative pain in adults. Cochrane Database Syst Rev. 2010 May 12;2010(5):CD008183. doi: 10.1002/14651858.CD008183.pub2. PMID 20464764
- [Background] Tiippana EM, Hamunen K, Kontinen VK, Kalso E. Do surgical patients benefit from perioperative gabapentin/pregabalin? A systematic review of efficacy and safety. Anesth Analg. 2007 Jun;104(6):1545-56, table of contents. doi: 10.1213/01.ane.0000261517.27532.80. PMID 17513656
- [Derived] Huynh TQ, Patel NR, Goldstein ND, Makai GE. Preoperative Gabapentin for Minimally Invasive Hysterectomy: A Randomized Controlled Trial. J Minim Invasive Gynecol. 2021 Feb;28(2):237-244.e2. doi: 10.1016/j.jmig.2020.04.040. Epub 2020 May 8. PMID 32389735

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient were recruited from June 2016 to July 2017 via phone or in the office setting. Potential subjects were informed of the study by investigators and if they desired to participate, they either signed consents forms in the office or on the day of surgery.
Pre-assignment Details: There were no events prior to assignment in study arm after participant enrollment.
Groups:
- Gabapentin: As per the enhanced recovery after surgery protocol at our health institution, subject will receive oral medications prior to surgery including acetaminophen, celecoxib, and gabapentin x 1 dose given preoperatively. The number of tablets and capsules will remain identical in both study arms. Medications given include:
  Gabapentin 600 mg (two capsules of gabapetin 300 mg); Acetaminophen 975 mg (three tablets of acetaminophen 325 mg); Celecoxib 400 mg (two capsules of celecoxib 200 mg) = Total 3 tablets, 4 capsules
  Gabapentin
  Acetaminophen
  Celecoxib
- Control: As per the enhanced recovery after surgery protocol at our health institution, subject will receive oral medications prior to surgery including acetaminophen and celecoxib x 1 dose given preoperatively. The number of tablets and capsules will remain identical in both study arms. Medications given include:
  Acetaminophen 975 mg (three tablets of acetaminophen 325 mg); Celecoxib 400 mg (four capsules of celecoxib 100 mg) = Total total 3 tablets, 4 capsules
  Acetaminophen
  Celecoxib
Period: 24 Hours Postoperative Assessment
Arm/Group | Gabapentin | Control
Started | 70 | 67
Completed | 68 | 61
Not Completed | 2 | 6
Not completed — Lost to Follow-up | 1 | 4
Not completed — excluded from analysis per protocol | 1 | 2
Period: 2 Weeks Postoperative Assessment
Arm/Group | Gabapentin | Control
Started | 68 | 61
Completed | 58 | 51
Not Completed | 10 | 10
Not completed — Lost to Follow-up | 10 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin | Control | Total
Number analyzed (Participants) | 68 | 61 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (12.56) | 52.3 (11.6) | 51.2 (12.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 61 | 129
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 43 | 46 | 89
  African American/African | 25 | 15 | 40
  Other | 1 | 4 | 5
Region of Enrollment [Number; unit: participants]
  United States | 68 | 61 | 129
BMI [Count of Participants; unit: Participants]
  < 30 kg/m^2 | 36 | 28 | 64
  >/= 30 kg/m^2 | 32 | 33 | 65
Narcotic Use within week prior to surgery [Count of Participants; unit: Participants] | 11 | 18 | 29
History chronic pain [Count of Participants; unit: Participants] | 26 | 24 | 50
Prior abdominal surgery [Count of Participants; unit: Participants] | 43 | 44 | 87
Preoperative pain score, within past week [Mean (Standard Deviation); unit: units on a scale] — Pain score assesses patient subjective pain via patient reported numeric analogue scale, range 0-10 with 0 being no pain and 10 being severe pain.
  units on a scale | 1.7 (2.9) | 2.0 (3.2) | 1.7 (3.0)
Preoperative pain score, within past 24 hours [Mean (Standard Deviation); unit: units on a scale] — Pain score assesses patient subjective pain via patient reported numeric analogue scale, range 0-10 with 0 being no pain and 10 being severe pain.
  units on a scale | 1.2 (2.5) | 1.1 (2.5) | 1.1 (2.5)
Preoperative pain score, in prep and hold [Mean (Standard Deviation); unit: units on a scale] — Pain score assesses patient subjective pain via patient reported numeric analogue scale, range 0-10 with 0 being no pain and 10 being severe pain.
  units on a scale | 1.0 (2.0) | 0.6 (1.4) | 0.7 (1.7)
Surgery Indication [Count of Participants; unit: Participants]
  Abnormal uterine bleeding | 31 | 21 | 52
  Leiomyomas | 28 | 18 | 46
  Adenomyosis | 1 | 2 | 3
  Pelvic pain | 15 | 18 | 33
  Endometriosis | 2 | 3 | 5
  Hyperplasia | 0 | 2 | 2
  Prolapse/Incontinence | 21 | 25 | 46
Hysterectomy Surgical Approach [Count of Participants; unit: Participants]
  Vaginal | 17 | 16 | 33
  Laparoscopic | 26 | 21 | 47
  Robotic | 25 | 24 | 49
Procedure other than Hysterectomy [Count of Participants; unit: Participants]
  Salpingectomy | 61 | 56 | 117
  Oophorectomy | 14 | 21 | 35
  Lysis of Adhesions | 9 | 5 | 14
  Sacral colpopexy | 7 | 6 | 13
  Sacropinous ligament fixation | 2 | 0 | 2
  Sling | 9 | 14 | 23
  Use of mesh | 11 | 15 | 26
  Cystoscopy | 48 | 49 | 97
  Uterosacral ligament fixation | 9 | 13 | 22
  Anterior/posterior repair | 9 | 12 | 21
  Paravaginal repair | 2 | 3 | 5
Method of specimen removal [Count of Participants; unit: Participants]
  Minilaparotomy | 10 | 5 | 15
  colpotomy | 56 | 56 | 112
  Power morcellation | 2 | 0 | 2
OR time [Mean (Standard Deviation); unit: minutes] | 186.3 (84.3) | 178.9 (74.6) | 183.8 (80.4)
Estimated blood loss [Mean (Standard Deviation); unit: mL] | 118.6 (106.6) | 155.9 (271.2) | 137.3 (206.9)

OUTCOME MEASURES:

1. Primary Outcome: Narcotic Use at 24 Hours Postop
Description: Assessment of the amount of narcotic use postoperatively at 24 hours. will use opioid equivalence table to convert all narcotic use to oxycodone equivalents
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: morphine milligram equivalents
Arm/Group | Gabapentin | Control
Number analyzed (Participants) | 68 | 61
morphine milligram equivalents | 158.8 (109.6) | 175.0 (162.5)

2. Primary Outcome: Subjective Pain at 24 Hours Postoperative
Description: Pain score assesses patient subjective pain via patient reported numeric analogue scale, range 0-10 with 0 being no pain and 10 being severe pain.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gabapentin | Control
Number analyzed (Participants) | 68 | 61
score on a scale | 3.4 (2.5) | 3.4 (2.5)

3. Secondary Outcome: Number of Patient With Gabapentin Adverse Effects at 24 Hours Postoperatively
Description: Will assess for known symptoms of gabapentin postoperatively at 24 hours. We will survey subjects regarding their experience of the following symptoms: dizziness/drowsiness, fatigue, loss of balance, blurry vision, tremulousness, swelling, nausea, vomiting, diarrhea, and allergic reaction
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Gabapentin | Control
Number analyzed (Participants) | 68 | 61
Participants
  Dizziness | 17 | 8
  Blurred Vision | 7 | 4
  Somnolence | 20 | 23
  Difficulty walking | 13 | 11
  Tremulousness | 11 | 6
  Nausea | 24 | 25
  Vomiting | 9 | 15

4. Secondary Outcome: Number of Patient With Gabapentin Adverse Effects at 2 Weeks Postoperatively
Description: Will assess for known symptoms of gabapentin postoperatively at 2 weeks. We will survey subjects regarding their experience of the following symptoms: dizziness/drowsiness, fatigue, loss of balance, blurry vision, tremulousness, swelling, nausea, vomiting, diarrhea, and allergic reaction
Time Frame: 2 weeks
Population: participants included in analysis differs from participant flow due to subjects loss to follow up at the 2 weeks time frame. study powered to primary outcome at 24 hours postoperative. 10 subjects were lost to follow up at 2 weeks postoperative in both the gabapentin and control arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Gabapentin | Control
Number analyzed (Participants) | 58 | 51
Participants
  Dizziness | 12 | 8
  Blurred vision | 4 | 3
  Somnolence | 18 | 21
  Difficulty walking | 5 | 5
  Tremulousness | 4 | 2
  Nausea | 12 | 7
  Vomiting | 0 | 1

5. Secondary Outcome: Narcotic Use at 2 Weeks Postop
Description: Assessment of the amount of narcotic use postoperatively at 2 weeks. will use opioid equivalence table to convert all narcotic use to oxycodone equivalents
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: morphine milligram equivalents
Arm/Group | Gabapentin | Control
Number analyzed (Participants) | 58 | 51
morphine milligram equivalents | 167.2 (79.3) | 187.3 (185.5)

6. Secondary Outcome: Subjective Pain at 2 Weeks Postop
Description: Assessment of the subject pain score postoperatively at 2 weeks. will use a numeric analog scale from 0-10.
  The pain scale ranging from 0-10 with 0 representing No Pain and 10 representing the Worst Pain Possible
Time Frame: 2 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gabapentin | Control
Number analyzed (Participants) | 58 | 51
score on a scale | 1.3 (2.0) | 1.4 (1.8)

ADVERSE EVENTS:
Time Frame: Adverse event data collected from time of enrollment to 2 weeks postoperative.
Arm/Group | Gabapentin | Control
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/67
Other Adverse Events (participants affected / at risk) | 0/70 | 0/67

LIMITATIONS AND CAVEATS:
Study limited by recall bias and imperfect patient blinding inherent in placebo equivalent methadology. Most patients discharged prior to 24 hours, therefore data collected dependent on patient reporting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-12): https://cdn.clinicaltrials.gov/large-docs/59/NCT02703259/Prot_SAP_000.pdf